CLINICAL TRIAL: NCT07070492
Title: Outcomes of Combined Cataract Surgery With Retinal Surgery for Visually Significant Epiretinal Membrane With Vivity Versus Monofocal Intraocular Lens
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Debbie Kuo, MD (Other)
Responsible Party: Sponsor-Investigator, Debbie Kuo, MD, Palo Alto Foundation Medical Group affiliated Ophthalmologist, Sutter Health
Organization: Sutter Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025.067-1
Record Dates: First submitted 2025-06-24; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cataract and IOL Surgery; Epi-retinal Membrane
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vivity Extended Depth of Focus IOL (Experimental)
  Interventions: Device: cataract surgery; Procedure: retinal surgery
- Standard monofocal IOL (Active Comparator)
  Interventions: Device: cataract surgery; Procedure: retinal surgery

INTERVENTIONS:
Device: cataract surgery — cataract surgery receiving Vivity IOL or standard mono focal controls
Procedure: retinal surgery — Retinal surgery for visually significant epiretinal membrane

SUMMARY:
To investigate the patient Quality of Life and satisfaction outcomes of combined cataract surgery with retinal surgery for visually significant epiretinal membrane in patients receiving Vivity IOL versus standard monofocal controls.

DETAILED DESCRIPTION:
The information gained by this study will help understand better the suitability of Vivity IOLs for patients with a common retinal condition and potentially expand access and offering of premium IOLs to help patients gain independence from glasses, which can improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with visually significant epiretinal membrane who are undergoing or have already had pars plana vitrectomy and membrane peel combined with cataract surgery using Clareon Vivity and Clareon Vivity Toric IOLs or monofocal IOL
* IOL powers between +6D to +30.0D, T3-T6

Exclusion Criteria:

* History of ocular or refractive surgery
* Other ocular or systemic comorbidities that may alter or reduce visual acuity and contrast sensitivity, such as severe dry eye/ocular surface disease, glaucoma, macular degeneration, retinopathy, neuro-ophthalmic diseases, strabismus/amblyopia etc.
* Patients with irregular astigmatism, corneal dystrophies, pupil abnormalities, zonular laxity
* Intraoperative or postoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Vision Acuity | At the study visit at least 3 months after the combined cataract and retinal surgeries

SECONDARY OUTCOMES:
Contrast Sensitivity | At the study visit at least 3 months after the combined cataract and retinal surgeries
Patient Reported Outcomes (PRO) on vision-related Quality of Life (QOL) and satisfaction | At the study visit at least 3 months after the combined cataract and retinal surgeries
  Using 5-point Likert scale, Research Insight's Validated PRO Questionnaire to assess patient overall satisfaction post-surgery, QOL on driving, reading, computer use, watching TV, sports, and Glare/Haloes.

IPD SHARING:
Plan to Share IPD: Yes
Patient Report Outcomes on Quality of Life and satisfaction
Supporting Information: SAP, CSR
Time Frame: After the final results were published and released to the public.
Access Criteria: Researchers will have to make explicit request to the corresponding author to determine if any individual participant data can be released. No Personal Health Information and personal identifiers will be shared.